CLINICAL TRIAL: NCT02570867
Title: Study on the Changes of Brain Function in Primary Open-angle Glaucoma Patients With fMRI
Brief Title: Functional Brain Changes of Primary Open-angle Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qing Zhou (Other)
Responsible Party: Sponsor-Investigator, Qing Zhou, Vice director of Department of Ophthalmology The First Affiliated Hospital of Jinan University, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: FirstJinanU
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Glaucoma
Keywords: glaucoma; brain function; fMRI
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal control group: Normal control group: healthy volunteers will be received Functional magnetic resonance imaging（fMRI) and eye examination including visual acuity, visual field, intraocular pressure, anterior chamber angle, corneal thickness and optic nerve fiber thickness one time.
- POAG group: POAG: The primary open angle glaucoma cases were will be received Functional magnetic resonance imaging（fMRI) and eye examination including visual acuity, visual field, intraocular pressure, anterior chamber angle, corneal thickness and optic nerve fiber thickness one time.

SUMMARY:
Structural and functional brain changes of primary open-angle glaucoma patient will be examined with fMRI. POAG patients and control group were examined with 3.0T magnetic resonance imaging. The gray matter, white matter and cerebrospinal fluid volume images will be obtained and analysed.

DETAILED DESCRIPTION:
More and more researches showed that nerve damage in glaucoma is not limited in the optic nerve, but also involved the visual pathway, including the optic chiasm, optic beam, lateral geniculate body, optic radiation and visual cortex. Furthermore, the central nervous system changes may be earlier than visual field and the optic nerve morphology change. Tomography (OCT), laser polarimetry 0ptical (SLP), evoked potential scanning (VEP) can not accurately reflect the central nervous system changes caused by glaucoma.

In recent years, magnetic resonance diffusion tensor imaging (DTI), blood oxygen level dependent functional magnetic resonance imaging(fMRI- BOLD) and voxel-based Morphometry（VBM) is widely used in clinical practice. The differences in the density and volume of brain tissue could be analyzed with VBM which had the advantages of comprehensive, objective and repeatable. Studies have indicated that patients with POAG can lead to a wide range of changes in the cerebral cortex which are associated with the severity of glaucoma.

Participants in the study will be assigned to primary open-angle glaucoma (POAG) patients or healthy volunteers. Two groups will be received 3.0T functional magnetic resonance imaging（fMRI) and eye examination including visual acuity, visual field, intraocular pressure, anterior chamber angle, corneal thickness and optic nerve fiber thickness. We hope this trial will reveal the patterns and structural differences of brain function abnormalities between the POAG patents and the normal people. And the same time, the correlation between brain gray changes and visual field and retinal nerve fiber layer thickness will be analysed.

ELIGIBILITY:
Inclusion Criteria（POAG patients）

1. ages of 18 and 40 years.
2. glaucoma diagnostic criteria: a) intraocular pressure(IOP) ≥ 21mmhg; b) glaucoma specific changes of optic papilla and retinal nerve fiber layer defect;c) glaucoma specific visual field defect; d) the anterior chamber angles are open.
3. without other eye diseases.
4. Written informed consent.

Inclusion Criteria（Healthy Volunteers）:

1. ages of 18 and 40 years.
2. eye examinations of best corrected visual acuity ≥20/20.
3. the equivalent degree of myopia < -6.00d.
4. IOP < 21 mmHg.
5. without other eye diseases;
6. Written informed consent.

Exclusion Criteria（POAG patients and Healthy Volunteers）:

1. ages over 40 years or less than 18 years.
2. myopic degree (equivalent refraction) is greater than 6.0D.
3. history of ocular trauma and ocular surgery.
4. with other eye diseases: corneal diseases, cataract, diabetic retinopathy and optic nerve diseases.
5. brain injury and other diseases of the nervous system: Alzheimer's disease, Parkinson's disease.
6. MRI scan showed that there was a qualitative change: cerebral infarction, cerebral thrombosis, etc.
7. install cardiac pacemakers, claustrophobic patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: POAG group :20 cases normal control group:20 cases
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes of Brain Function | 18 months
  The gray matter, white matter and cerebrospinal fluid volume images will be obtained with 3.0T magnetic resonance imaging. The two groups will be compared by Two Sample T-Test.

SECONDARY OUTCOMES:
Correlation between brain gray changes and retinal nerve fiber layer thickness | 18 months
  Brain grey matter volume will be measured with 3.0T magnetic resonance imaging and the optic nerve fiber layer thickness were measured with OCT. The correlation of the two will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhou, MD, Study Chair — First Affiliated Hospital of Jinan University; Qing Zhou, MD, Principal Investigator — First Affiliated Hospital of Jinan University
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Background] He M, Foster PJ, Ge J, Huang W, Zheng Y, Friedman DS, Lee PS, Khaw PT. Prevalence and clinical characteristics of glaucoma in adult Chinese: a population-based study in Liwan District, Guangzhou. Invest Ophthalmol Vis Sci. 2006 Jul;47(7):2782-8. doi: 10.1167/iovs.06-0051. PMID 16799014
- [Background] Gupta N, Yucel YH. What changes can we expect in the brain of glaucoma patients? Surv Ophthalmol. 2007 Nov;52 Suppl 2:S122-6. doi: 10.1016/j.survophthal.2007.08.006. PMID 17998036
- [Background] Ito Y, Shimazawa M, Chen YN, Tsuruma K, Yamashima T, Araie M, Hara H. Morphological changes in the visual pathway induced by experimental glaucoma in Japanese monkeys. Exp Eye Res. 2009 Aug;89(2):246-55. doi: 10.1016/j.exer.2009.03.013. Epub 2009 Mar 31. PMID 19341728
- [Background] Gupta N, Ang LC, Noel de Tilly L, Bidaisee L, Yucel YH. Human glaucoma and neural degeneration in intracranial optic nerve, lateral geniculate nucleus, and visual cortex. Br J Ophthalmol. 2006 Jun;90(6):674-8. doi: 10.1136/bjo.2005.086769. Epub 2006 Feb 7. PMID 16464969
- [Background] Murai H, Suzuki Y, Kiyosawa M, Tokumaru AM, Ishii K, Mochizuki M. Positive correlation between the degree of visual field defect and optic radiation damage in glaucoma patients. Jpn J Ophthalmol. 2013 May;57(3):257-62. doi: 10.1007/s10384-013-0233-0. Epub 2013 Feb 16. PMID 23417328
- [Background] Qing G, Zhang S, Wang B, Wang N. Functional MRI signal changes in primary visual cortex corresponding to the central normal visual field of patients with primary open-angle glaucoma. Invest Ophthalmol Vis Sci. 2010 Sep;51(9):4627-34. doi: 10.1167/iovs.09-4834. Epub 2010 Mar 31. PMID 20357191
- [Background] Chen WW, Wang N, Cai S, Fang Z, Yu M, Wu Q, Tang L, Guo B, Feng Y, Jonas JB, Chen X, Liu X, Gong Q. Structural brain abnormalities in patients with primary open-angle glaucoma: a study with 3T MR imaging. Invest Ophthalmol Vis Sci. 2013 Jan 17;54(1):545-54. doi: 10.1167/iovs.12-9893. PMID 23258150
- [Derived] Jiang MM, Zhou Q, Liu XY, Shi CZ, Chen J, Huang XH. Structural and functional brain changes in early- and mid-stage primary open-angle glaucoma using voxel-based morphometry and functional magnetic resonance imaging. Medicine (Baltimore). 2017 Mar;96(9):e6139. doi: 10.1097/MD.0000000000006139. PMID 28248867